CLINICAL TRIAL: NCT05789420
Title: A Single-center, Randomized, Controlled, Open-label Study in Smoking Healthy Subjects to Investigate the Nicotine Pharmacokinetic Profiles Following Single Use of Tobacco Heating System (THS) With a Regular or a Menthol Stick, Compared to Smoking of a Single Combustible Cigarette (CIG)
Brief Title: Nicotine Pharmacokinetics of THS Single Use of a Regular or a Menthol Stick Compared to CIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P1-PK-12
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Smoking, Tobacco
Keywords: Nicotine; Nicotine-containing products; Heated tobacco; Smoking; Tobacco; Tobacco Heating System; Pharmacokinetics
MeSH Terms: conditions — Tobacco Smoking; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product Sequence 1 (Active Comparator): After at least 23 hours of abstinence from any Tobacco or Nicotine Product (TNP) on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or performed a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG
- Product Sequence 2 (Active Comparator): After at least 23 hours of abstinence from any TNP on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or performed a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG
- Product Sequence 3 (Active Comparator): After at least 23 hours of abstinence from any TNP on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or performed a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG
- Product Sequence 4 (Active Comparator): After at least 23 hours of abstinence from any TNP on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or performed a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG
- Product Sequence 5 (Active Comparator): After at least 23 hours of abstinence from any TNP on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or perform a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG
- Product Sequence 6 (Active Comparator): After at least 23 hours of abstinence from any TNP on Day 1, and after at least 23 hrs of former IP use on Day 2 and Day 3 (nicotine wash-out), subjects smoked a single CIG or perform a single use of a THS either with a regular or a menthol THS stick, according to randomized product use sequence.
  The list of possible sequences are:
  P1R; P1M; CIG / P1R; CIG; P1M / P1M; P1R; CIG / P1M; CIG; P1R / CIG; P1R; P1M / CIG; P1M; P1R
  Interventions: Other: P1R stick; Other: P1M stick; Other: CIG

INTERVENTIONS:
Other: P1R stick — Regular flavor tobacco stick
Other: P1M stick — Mentholated flavor tobacco stick
Other: CIG — Subjects' preferred brand of commercially available, regular or mentholated cigarettes

SUMMARY:
The purpose of this study was to describe the nicotine pharmacokinetic (PK) profile during and after single use of THS (Induction heating technology, with either a regular or menthol stick) compared to singular CIG smoking in healthy adult subjects. In addition, pharmacodynamic effects (subjective effects) were evaluated to provide further insights on product acceptance and likelihood to use the THS again. Safety was assessed throughout the study.

DETAILED DESCRIPTION:
General information about the research:

Study Title:

Nicotine Pharmacokinetics of THS Single Use of a Regular or a Menthol Stick Compared to CIG

Who carried out the research? This research was sponsored and funded by Philip Morris Products S.A.

What public involvement there was in the study? Thirty-one healthy, currently smoking, adults participated in this study.

Where and when the study took place? The study was conducted at a clinical trial facility managed by a contract research organization in Belfast, Northern Ireland, from February 16th to April 2nd 2023.

Why was the research needed? The research was needed to understand the nicotine pharmacokinetic profile of the Tobacco Heating System (THS), with induction heating technology, in healthy smokers following single use of THS, with a regular or menthol stick, compared to cigarette single-use.

What were the main questions studied? The study measured the amount and the time rate of nicotine uptake in blood plasma, and other parameters. These were the maximum nicotine plasma concentration [Cmax], the time to the maximum nicotine plasma concentration [Tmax], and further subsequent calculations describing the nicotine exposure profile.

Who participated in the study? Thirty-one healthy, male or female, adults aged between 21 and 65 years participated in this study. All participants were currently smoking. The participants did not plan to quit using tobacco and/or nicotine products within the next 3 months and had smoked continuously for at least the last 3 years prior to joining the study.

Each participant was given full and adequate oral and written information about the nature, purpose, possible risks, and benefits of the study.

All participants received information on the risks of smoking, smoking cessation advice and a briefing on the Tobacco Heating System, for example, that its use is not risk-free.

Once each participant had received all the necessary information, and if they agreed to participate, this was documented in an Informed Consent Form with the date, time, and signature of both the participant and the study doctor.

Participants were informed that they were free to withdraw from the study at any time.

What treatments or interventions did the participants take/receive? Thirty participants were randomly assigned to one of six possible cross-over sequences of product use (THS, with either regular or menthol stick, and cigarette) from Day 1 to Day 3 in a confinement setting.

Participants could not use any other tobacco or nicotine-containing product (TNP) other than their assigned product.

From Day 1 to Day 3, after at least 23 hours of abstinence from any TNP on Day 1, and at least 24 hours after former IP use on Day 2 and on Day 3 (nicotine washout), subjects smoked a CIG or used the THS either with a regular or a menthol THS stick according to their randomized product use sequence.

Blood samples were collected, at several time points after product use, from Day1 to Day 3, for determination of nicotine concentration after allocated product use.

Participants were also asked, from Day 1 to Day 3, to evaluate product liking, craving for cigarettes, and their intention to use the product again. These were assessed on a scale for each evaluation. The scales went from "strong disliking" to "strong liking" for product liking; from "no craving" to "strong craving" for cigarette craving; and "very unlikely" to "very likely" for intention to use again.

What medical problems (adverse reactions) did the participants have? Overall, there were six mild adverse reactions reported in four participants. All the adverse reactions were mild or moderate in severity. None of these were considered related to an investigational product.

There were no clinically significant findings in the physical examination, clinical laboratory, vital signs, or ECG assessments in this study.

What happened during the study? A presentation of THS (without product use) was made to the participants during the Screening visit. All participants received information on the risks of smoking, smoking cessation advice, and a briefing that the use of THS is not risk-free.

Eligible participants, fulfilling all criteria for participation, returned to the investigational site for admission and baseline measurements on Day -1.

Subjects fasted for at least 6 hours prior to the safety laboratory assessments and started abstinence of TNP.

Thirty subjects were randomized to one of 6 possible full cross-over sequences of product use (THS, with either regular or menthol THS stick, and cigarette) on Day 1 to Day 3.

On Day 1 to Day 3, after at least 23 hours of abstinence from any TNP on Day 1, and at least 24 hours after THS use on Day 2 and on Day 3 (nicotine washout), subjects smoked a cigarette or used the THS either with a regular or a menthol THS stick according to randomized product use sequence.

Blood samples were obtained according to the standard procedures of the investigational site. Subjects were requested to report their cigarette craving, THS liking, and intention to use the THS again.

After Discharge on Day 3 or after an early termination following product exposure, the subjects entered a 3-day Safety Follow-Up period during which adverse reactions reported by the subjects were collected and followed-up, concluded by telephone contact by the investigational site on the last day of the Safety Follow-Up period.

What were the results of the study? The nicotine exposure profiles and subjective effects of THS product use were assessed for THS tobacco sticks of different flavors (regular flavor; menthol flavor) and compared to those of cigarette smoking.

The results of this study confirmed that nicotine exposure, from both THS Regular tobacco sticks and THS Menthol tobacco sticks, showed a lower level of nicotine uptake when using the THS Induction device compared to cigarette single use. These results are in line with historical data described for the THS device with blade heating technology.

The subjective effects of THS (induction) use were comparable to those presented in previous studies that compared THS (blade) use to cigarette use, which found that cigarette use was more satisfying while THS demonstrated comparable craving reduction.

Furthermore, this study found no additional safety concerns were associated with THS compared to cigarette smoking.

How has this study helped patients and researchers? The participants in this study were healthy, current cigarette smokers. All participants were informed about the health risks associated with smoking and were given smoking cessation advice. Participants in this clinical study benefited from repeated and detailed general health check-ups.

This clinical study may help doctors and scientists learn about electronic nicotine delivery systems.

Details of any further research planned This study is part of an ongoing program of research supporting the scientific substantiation of the Tobacco Heating System.

Where can I learn more about this study?

More details about this study, including the study results and a copy of the study protocol, can be found on the clinicaltrials.gov website at this address:

https://clinicaltrials.gov/show/NCT05789420

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the ICF and is able to understand the information provided in the ICF.
* Subject has been a smoker for ≥3 years prior to the screening visit (smoking cessation attempts during this period, if any, did not last > 6 months in total).
* Subject has continuously smoked on average ≥10 commercially available regular CIG/day over the last 4 weeks. Smoking status will be verified based on a urinary cotinine test (cotinine ≥200 ng/mL).
* Subject is healthy as judged by the Investigator based on available assessments from the screening period (e.g., safety laboratory, spirometry, vital signs, physical examination, ECG, and medical history).
* Subject does not plan to quit smoking within the next three months.

Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason other than medical (e.g., psychological, social reason).
* Subject is legally incompetent, or physically or mentally incapable of giving consent (e.g., in emergency situations, under guardianship, prisoners).
* Subject has a clinically relevant disease which requires medication (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, oncological, urological, immunological, pulmonary, and cardiovascular disease) or any other medical condition (including safety laboratory), which as per the judgment of the Investigator would jeopardize the safety of the subject.
* Subject experienced within 30 days prior to screening/admission a body temperature >37.5°C or an acute illness (e.g., upper respiratory-tract infection, viral infection, etc.) or the subject has a confirmed or suspected active COVID-19 infection (based on the signs and symptoms observed at the time of assessment)
* As per the Investigator's judgment, the subject has medical conditions which do or will require a medical intervention (e.g., start of treatment, surgery, hospitalization) during the study participation, which may interfere with the study participation and/or study results.
* Subject has relevant history of, or current asthma condition or COPD condition, and/or clinically significant findings.
* Subject has donated blood or received whole blood or blood products within 3 months.
* BMI < 18.5 kg/m2 or ≥ 32.0 kg/m2.
* Positive serology test for HIV 1/2, HBV, or HCV.
* Subject has a positive alcohol breath test and/or has a history of alcohol disorder that could interfere with their participation in the study.
* The subject has a positive urine drug test.
* Subject or one of their family members is a current or former employee of the tobacco or e-cigarette industry.
* Subject or one of their family members is an employee of the investigational site or of any other parties involved in the study.
* Subject has participated in another clinical study within 3 months.
* Subject has been previously screened or enrolled in this study.
* Subject is pregnant (does not have negative pregnancy tests at Screening and at Baseline) or is breastfeeding.
* For women of childbearing potential only: subject does not agree to use an acceptable method of effective contraception.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-04-02 (Actual); Study Completion 2023-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Jaumont, MD, Study Chair — Philip Morris Products S.A.
Locations (1):
- Celerion, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 subjects were screened for the study who gave informed consent and had at least one safety assessment, which were the criteria for inclusion in the Safety Population. 31 subjects were enrolled (one subject completed alternate status but was not needed for study participation due to closed enrollment). One of the enrolled subjects was discontinued due to positive alcohol breath and urine tests on Day -1. A total of 30 subjects were randomized to participate in the study.
Groups:
- Safety Population: The safety population consisted of all subjects (screened [32], enrolled [31], and randomized [30]) who gave informed consent and had at least one safety assessment.
Period: Screening and Safety Assessments
Arm/Group | Safety Population
Started | 32
Completed | 31
Not Completed | 1
Not completed — Completed Alternate Status | 1
Period: Enrollment
Arm/Group | Safety Population
Started | 31
Completed | 31
Not Completed | 0
Period: Randomization to Product Assessments
Arm/Group | Safety Population
Started | 31
P1R Stick (Regular flavor tobacco stick) | 30
P1M Stick (Mentholated flavor tobacco stick) | 30
CIG (Subject's preferred brand of commercially available, regular or mentholated cigarettes) | 30
Completed | 30
Not Completed | 1
Not completed — Failed alcohol breath test and urine test on day -1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population.
Arm/Group | Safety Population
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (10.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 32
  Not Hispanic or Latino | 32
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 26.037 (2.8629)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration [Cmax]
Description: To measure Cmax from the single use of THS with either a regular or a menthol stick or of a single cigarette.
Time Frame: Measured from start of product use to 24 hours
Population: Some participants were excluded from analysis for protocol deviations (including, but not limited to, missing measurements).
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- P1R (THS Regular Stick): Randomized subjects exposed to P1R (THS Regular Stick).
- P1M (THS Menthol Stick): Randomized subjects exposed to P1M (THS Menthol stick).
- CIG (Cigarette): Randomized subjects using their own Cigarettes (CIG).
Arm/Group | P1R (THS Regular Stick) | P1M (THS Menthol Stick) | CIG (Cigarette)
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 8.425 [6.582 to 10.780] | 7.475 [5.464 to 10.23] | 13.43 [10.29 to 17.53]

2. Primary Outcome: Time to the Maximum Concentration [Tmax]
Description: To measure Tmax from the single use of THS with either a regular or a menthol stick or of a single cigarette.
Time Frame: Measured from start of product use to 24 hours
Measure: Median (Full Range); unit: minutes
Arm/Group | P1R (THS Regular Stick) | P1M (THS Menthol Stick) | CIG (Cigarette)
Number analyzed (Participants) | 30 | 30 | 30
minutes | 6.025 [3.73 to 32.3] | 5.942 [3.87 to 60.0] | 7.725 [5.93 to 30.0]

3. Primary Outcome: Area Under the Curve of Nicotine Plasma Concentration-time Computed From T0 to T=24 Hours [AUC0-24h]
Description: To measure AUC0-24h from the single use of THS with either a regular or a menthol stick or of a single cigarette.
Time Frame: Measured from start of product use to 24 hours
Measure: Geometric Mean (95% Confidence Interval); unit: ng*min/mL
Arm/Group | P1R (THS Regular Stick) | P1M (THS Menthol Stick) | CIG (Cigarette)
Number analyzed (Participants) | 30 | 30 | 30
ng*min/mL | 879.4 [682.1 to 1134] | 715.5 [510.0 to 1004] | 1436 [1085 to 1901]

4. Primary Outcome: Area Under the Curve of Nicotine Plasma Concentration-time Computed From T0 to the Subject-specific Time of Maximum Nicotine Concentration [AUC0-t']
Description: To measure the area under the curve of nicotine plasma concentration-time computed from T0 to the subject-specific time of maximum nicotine concentration [AUC0-t'], from the single use of THS with either a regular or a menthol stick or from a single cigarette. (AUC0-Tmax)
Time Frame: Measured from start of product use to 24 hours
Measure: Geometric Mean (95% Confidence Interval); unit: ng*min/mL)
Arm/Group | P1R (THS Regular Stick) | P1M (THS Menthol Stick) | CIG (Cigarette)
Number analyzed (Participants) | 30 | 30 | 30
ng*min/mL) | 40.16 [32.02 to 50.36] | 29.22 [22.08 to 38.66] | 58.23 [47.13 to 71.95]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 34 days.
Description: Adverse Events were collected for all subjects who gave informed consent and had at least one safety assessment, which included all screened (32 subjects), enrolled (31 subjects), and randomized (30 subjects).
Groups:
- Safety Population: The safety population consisted of all subjects (screened [32 subjects], enrolled [31 subjects], and randomized [30 subjects]) who gave informed consent and had at least one safety assessment.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

LIMITATIONS AND CAVEATS:
This was a single product use study, in which participants had no previous experience with the product. Therefore, it did not allow subjects to get familiar with the product.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/20/NCT05789420/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05789420/SAP_001.pdf